CLINICAL TRIAL: NCT00532207
Title: Efficacy and Safety of Teriparatide 20 Micrograms in the Treatment of Postmenopausal Women With Osteoporosis
Brief Title: Study of Teriparatide in the Treatment of Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8736; B3D-MW-GHCR
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Osteoporosis, Post-Menopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: teriparatide

INTERVENTIONS:
Drug: teriparatide — subcutaneous 20 micrograms
  Other Names: LY333334

SUMMARY:
To see if using teriparatide for 12 months will increase Bone Mineral Density at the lumbar spine in postmenopausal women with osteoporosis

ELIGIBILITY:
Inclusion Criteria:

* Are postmenopausal women at least 55 years old and at least 2 years postmenopausal at the time of entry into the trial, and who have given informed consent before entering the study and after being informed of the risks, medications, and procedures to be used in the study. In addition, women below the age of 60 years with indeterminate menopause due to premenopausal hysterectomy must have their postmenopausal status confirmed with a serum FSH level > 30 IU/L.
* Posterior-anterior lumbar spine (L1-L4) BMD and/or femoral neck BMD measurement at least < 2.5 standard deviation (SD) from the mean of healthy, pre-menopausal women.
* Results of lumbar BMD (L1-L4) measurement must be available. The initial lumbar spine assessment and the determination of the patient's eligibility for entry into the screening phase will be made by the individual investigator. If the L-1 vertebra cannot be analyzed due to artifact, vertebral fracture, osteophytes, or other abnormalities, that vertebra should be excluded from the analysis.
* Normal or clinically insignificant abnormal laboratory values (as defined by the investigator) including serum calcium, 25 hydroxyvitamin D levels and alkaline phosphatase.
* Willing to be trained on and use a pen type injection delivery system on a daily basis for 12 months.

Exclusion Criteria:

* Active liver disease - liver enzymes (ALT, AST) more than three times the upper normal range, or a bilirubin of > 2.0 mg/dl, or clinical jaundice.
* Abnormal thyroid function not corrected by therapy. Normal thyroid function will be documented by a normal TSH during screening phase
* History of active nephrolithiasis or urolithiasis in the prior 2 years. Patients with any documented history of nephro- or urolithiasis must have had an appropriate imaging procedure within the prior 6 months, such as, an intravenous pyelography (IVP), supine radiograph of the kidney ureter bladder (KUB), or renal ultrasound, which must document the absence of stones
* History of malignant neoplasms within the prior 5 years, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitively treated. If malignant neoplasm was ever diagnosed, patient must presently be free of disease.
* Current pharmacological treatment for osteoporosis, other than calcium and Vitamin D
* History of Paget's disease, renal osteodystrophy, osteomalacia, any secondary causes of osteoporosis, hyperparathyroidism (uncorrected), and intestinal malabsorption

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-11; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that therapy for 12 months with once daily subcutaneous PTH 1-34 (teriparatide; TPTD) 20 micrograms will increase Bone Mineral Density (BMD) at the lumbar spine in postmenopausal women with osteoporosis

SECONDARY OUTCOMES:
To test the hypothesis that therapy for 3 months with once daily subcutaneous teriparatide 20 micrograms will increase markers of bone formation (P1NP, BSAP) and bone resorption (serum CTX) in postmenopausal women with osteoporosis
To test the hypothesis that therapy for 12 months with once daily subcutaneous teriparatide 20 micrograms will increase markers of bone formation (P1NP, BSAP) and bone resorption (serum CTX) in postmenopausal women with osteoporosis.
To evaluate safety of once daily subcutaneous teriparatide 20 micrograms for 12 months.
To evaluate effect of teriparatide on changing in femoral neck and total hip BMD
To test the hypothesis that treatment with TPTD will favorably affect back pain within the natural course of the disease
To test the hypothesis that treatment with TPTD will favorably affect quality of life within the natural course of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow, Russia

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com